CLINICAL TRIAL: NCT01993004
Title: Immune Regulation in Multiple Sclerosis: The Effect of Glatiramer Acetate on MicroRNA Expression in Antigen-Presenting Cells
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Konstantin Balashov, Associate Professor, Rutgers, The State University of New Jersey
Other Study IDs: IRB0220060134
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy subjects: Self-explanatory
- Untreated patients: Patients diagnosed with relapsing-remitting multiple sclerosis (RRMS) or clinically isolated syndrome (CIS) who are not on any disease-modifying treatment approved for MS
- Treated patients: Patients diagnosed with relapsing-remitting multiple sclerosis (RRMS) or clinically isolated syndrome (CIS) who were prescribed Glatiramer acetate prior to enrollment

SUMMARY:
MicroRNAs regulate gene expression. The abnormal expression of microRNAs has been reported in many human diseases. The purpose of this pilot study is to determine if microRNA expression is changed in untreated and glatiramer acetate-treated patients with multiple sclerosis.

DETAILED DESCRIPTION:
MicroRNAs regulate gene expression. The abnormal expression of microRNAs has been reported in many human diseases. The purpose of this pilot study is to determine if microRNA expression is changed in untreated and glatiramer acetate-treated patients with multiple sclerosis. The expression of microRNA will be analysed in cell subsets separated from peripheral blood mononuclear cells.

ELIGIBILITY:
Inclusion Criteria:

18-60 year-old healthy subjects or patients with RRMS/CIS

Exclusion Criteria:

1. Any treatment with steroids in the last 30 days prior to the blood draw or any immunosuppressive or Disease-modifying treatment (DMT) other than Glatiramer Acetate in the last 90 days
2. Presence of other disorders that may be associated with immune-deficient or autoimmune process (e.g., HIV, lymphoma, lupus) or demyelinating disease other than MS (e.g., Lyme, B12 deficiency)
3. Pregnancy
4. Intermittent or unilateral constant assistance (cane, crutch, brace) required to walk about 100 meters with or without resting (Expanded Disability Status Scale (EDSS) score greater than 5.5)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Control human subjects and patients with RRMS will be enrolled in New Brunswick, NJ
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Relative MicroRNA expression in B cells | 1 day
  Expression of multiple microRNA is being tested in B cells in three groups of subjects at one time point

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin Balashov, MD, PhD, FAAN, Principal Investigator — Rutgers-RWJMS
Locations (1):
- Rutgers-RWJMS, New Brunswick, New Jersey, United States